CLINICAL TRIAL: NCT05061225
Title: The Efficacy of a Facebook-delivered Physical Activity Counselling Intervention on Mental Health in Firefighters: a Randomized Controlled Trial
Brief Title: The Efficacy of a Physical Activity Counselling Intervention on Mental Health in Firefighters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Collaborators: Fire Stress Team (Unknown)
Responsible Party: Principal Investigator, Davy Vancampfort, Prof. dr., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3M200373
Record Dates: First submitted 2021-09-03; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: PTSD; Stress, Psychological; Depressive Symptoms; Anxiety Disorders and Symptoms
Keywords: Exercise; PTSD; Firefighter; Physical Activity; Stress; Depression; Anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress, Psychological; Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants invited to the private Facebook group
  Interventions: Behavioral: Physical activity counselling
- Waiting list (No Intervention): Waiting list. Will be invited to Facebook group after finalising the study and will receive same intervention.

INTERVENTIONS:
Behavioral: Physical activity counselling — Educational content on several topics regarding physical activity and its implementation in daily living
  Arms: Intervention

SUMMARY:
Objectives: The aim of this project will be to evaluate the efficacy of a lifestyle PA counselling program for physically inactive first responders with at least mild symptoms of either anxiety, depression or stress and their chosen support partners compared to a waiting list, and to determine the mediating effect of autonomous motivation. Additionally, the randomised controlled trial will be complemented with qualitative interviews to provide a deeper context and understanding to the quantitative findings. To the best of our knowledge, no randomized controlled trial to date has examined the outcomes of an online physical activity counselling intervention using peer-support in firefighters.

Methods: Within mixed methods randomized controlled trials, we will follow a sequential explanatory design. In this design, qualitative results complement and help interpret quantitative findings. In order to address the main aims, a randomized controlled trial will be executed. CONSORT statement will be followed for reporting findings. Protocol will be submitted to clinicaltrials.gov. For addressing the secondary aim of the study, the study will follow a qualitative design based on interpretative phenomenology. Phenomenology is a model used for describing, understanding, and interpreting the lived experiences of the participants by means of discourse analysis. For the quantitative component, two arms with 24 firefighters will be required. Additionally, chosen support partners will enter the intervention arm. Participants in the intervention arm will be invited to a private facebook page where the researcher will upload weekly educational posts regarding different aspects of physical activity. For the qualitative component, participants will be invited to 2-3 focus groups where the experiences of the participants on the program will be discussed.

DETAILED DESCRIPTION:
Background:

Posttraumatic stress disorder (PTSD) is characterized by a combination of emotional, behavioural, and physiological symptoms following exposure to a traumatic event. Due to a greater exposure to traumatic events, first responders such as firefighters tend to have worse general well-being, higher risk of problematic alcohol use, and worse sleep quality, which consequently results in mental health problems, and also increases the risk of firefighters of developing PTSD compared to the general population. Evidence-based guidelines for the treatment of PTSD consider psychotherapy and pharmacotherapy as first line treatment. However, less than 10% of first responders with PTSD seek these guideline-informed treatments. One of the reasons is that first responders have a unique culture of self-reliance and strength, where mental health issues are considered a weakness. A culture of not showing weakness, together with fear of stigma and of confidentiality breach are the main barriers for seeking traditional mental health treatment.

Physical activity (PA) and its structured form, exercise, are a non-stigmatizing, easily accessible and promising add-on prevention and treatment interventions for a wide range of mental disorders including depression, anxiety- and stress-related disorders. It has an effect size similar to commonly used pharmacotherapy in patients with anxiety disorders. Furthermore, PA-based interventions have shown to be effective in improving sleep quality and reducing alcohol consumption. Adding on the mental health benefits, PA-based interventions can also target the cardiometabolic co-morbidity commonly observed in people with depression, anxiety- and stress-related disorders and in first responders. Therefore, PA might be a promising treatment modality for physically inactive first responders with depression, anxiety, or stress symptoms. Current guidelines strongly recommend 150-300 minutes of moderate PA or 75-150 minutes of vigorous PA, or an equivalent combination of moderate-to-vigorous PA.

In order to successfully implement PA-based interventions as prevention and treatment programs, research should explore effective ways to deliver the intervention in a way that is appealing for the target population. E-health and new technologies could provide a novel and less stigmatising approach to mental health interventions. It is an accessible and low-cost tool that could be effective for delivering PA interventions, increasing PA levels and improving mental health outcomes in people with psychiatric disorders or mental distress. Social media, more specifically Facebook, is a promising platform that has been previously used for supporting PA interventions for people with severe mental illness. The use of a private Facebook group to deliver these interventions could increase the feeling of belongingness and facilitate peer-to-peer support.

Social support is an essential aspect of adherence to PA interventions. Furthermore, social and family support are well-known protective factors against mental distress after prolonged exposure to trauma. Recent research suggests that partners, family members, or friends (commonly known as "informal caregivers") of first responders with mental distress have poorer mental health compared with the general population. Moreover, informal caregivers are also more likely to be sedentary, defined as wake-time spent sitting, reclined, or lying down quietly, than the general population. Including informal caregivers as support partners in a PA intervention could be beneficial not only for the first responders, but for the health of their informal caregivers. Another relevant factor which has been found to impact implementation of PA in daily living is the quality of the motivation to engage in PA. Previous research has found evidence that higher levels of autonomous motivation are related to more leisure time spent in physical activity in firefighters. However, despite the calls for more research examining the mediating effect of autonomous motivation on PA-based interventions, there is still a lack of causal evidence on the influence of autonomous motivation on PA-related behaviour change in physically inactive firefighters.

Therefore, the aim of this project will be to evaluate the efficacy of a lifestyle PA counselling program for physically inactive first responders with at least mild symptoms of either anxiety, depression or stress and their chosen support partners compared to a waiting list, and to determine the mediating effect of autonomous motivation. Additionally, the randomised controlled trial will be complemented with qualitative interviews to provide a deeper context and understanding to the quantitative findings. To the best of our knowledge, no randomized controlled trial to date has examined the outcomes of an online physical activity counselling intervention using peer-support in firefighters.

Aims:

Main aims:

• To evaluate the efficacy of a lifestyle PA counselling program in physically inactive firefighters with depression, anxiety and stress symptoms and their support partner compared to waiting list.

Secondary aims:

* To evaluate the mediating effect of autonomous motivation and perceived social support on the improvements on PA levels and mental health outcomes after a lifestyle PA counselling program.
* To understand the experiences of firefighters and their support partners participating in a lifestyle PA counselling program.

General hypotheses

Based upon of the aforementioned aims, the following hypotheses will be tested:

* PA levels, mental health outcomes, quality of life, and sleep quality of firefighters and their support partners will improve after participating in a PA counselling intervention.
* Autonomous motivation and perceived social support will partially mediate the improvements on PA levels and mental health outcomes of firefighters after participating in a PA counselling intervention.

It is important to indicate that qualitative research does not require a hypothesis, but a research question to drive the study. The research question for the secondary aim of the study is "How is the experience of participating in a PA counselling intervention to increase levels of PA and improve mental health outcomes, quality of life and sleep quality?".

Design:

Mixed-methods designs facilitate the assessment of the perspectives and experiences of the participants while providing numerical data, and can offer deeper and wider understanding of a research question than qualitative or quantitative methodologies alone. For this reason, the use of mixed-methods designs in mental health research and implementation of new health policies is growing. Furthermore, this design is recommended for physical therapy and rehabilitation research aimed at exploring and explaining complex phenomena in interaction with bio-psycho-social and personal factors. This study will explore the complexity of the interactions between motivation for PA, mental health, and traumatic experiences for which the use of a purely quantitative or qualitative approach would be insufficient.

Within mixed methods randomized controlled trials, a sequential explanatory design will be followed. In this design, qualitative results complement and help interpret quantitative findings. In order to address the main aims, a randomized controlled trial will be executed. CONSORT statement will be followed for reporting findings. Protocol will be submitted to clinicaltrials.gov. For addressing the secondary aim of the study, the study will follow a qualitative design based on interpretative phenomenology. Phenomenology is a model used for describing, understanding, and interpreting the lived experiences of the participants by means of discourse analysis.

Methods:

Members of Fire Stress Team (FiST) will be contacted, a non-profit community initiative aiming to increase awareness for support and care for first responders and their families, and Netwerk Brandweer Vlaanderen, the firefighters' network of the Flemish region of Belgium. Participants will be recruited via mail in which they will receive the participant information and a flyer of the study. Participants will have the option to schedule a meeting with the main researcher to go through possible questions or comments.

Participants should have internet access and an active Facebook account or be willing to create one. First-responders will be required to nominate a support partner. This may be any person with a close personal relationship to them, for example, partner, family member, carer or friend with whom they have at least weekly in-person contact with. Participants who are eligible will be randomized to either the lifestyle PA counselling or a wait-list condition.

To avoid separating firefighters from their support partner, each pair will be randomized as a unit. Each group will have the same number of participants (1:1). Each pair will be coded by a research assistant, who will do the simple randomization into control or intervention arm before baseline assessment using www.randomization.com. Allocation will be concealed from participants and the main researcher. The research assistant will introduce the allocation results in a sealed opaque envelope which will only be opened once baselines assessments have been completed in order to invite the participants to the Facebook group.

G*Power was used to detect an average large effect size (r = 0.8) with a statistical power of 80% and a significance level of 0.05 based on the SD of a similar population. A total sample size of 24 firefighters per group for each intervention study is required to detect a 10 point between group difference on the PCL-5. An additional number of 6 firefighters will be recruited to account for a possible drop-out rate of 22% based on the results of the latest literature on drop-out rates on exercise trials for anxiety and related- disorders.

Assessments will be executed on 3 time points for both intervention and control group: one-week pre- intervention, immediately post- intervention and 3 months post. The full survey takes approximately 50 minutes to complete. Data will be stored separately for control and intervention arm. A survey with all the questionnaires will be sent by e-mail to the participants. Blinding at baseline will be reached by concealed allocation, and a researcher blinded to group allocation will carry out assessments post-intervention and at 3-month follow-up.

The PA counselling intervention will consist of 10 weeks of content, delivered online interventions through a private Facebook page. Firefighters and their nominated support partners will both be encouraged to be actively involved on the Facebook page and with the programme. The research team will facilitate discussion boards. The intervention will be elaborated based on the evidence gathered in previous studies on the different motivation strategies and barriers for PA. Weekly content will include information regarding different aspects of physical activity and mental health, demonstration videos, links to existing online resources and discussion questions. These posts will all occur from the study generated account, twice a week, and the page will be checked by the researcher at least once per day, Monday to Friday. If participants are not interacting (i.e. reading the posts) in the Facebook page for more than a week they will be contacted by the main researcher. At the beginning of the intervention, participants will be given a Fitbit Inspire 2 in order to learn self-monitoring and goal-setting. An outline of the intervention content can be found in Table 1. Behaviour-change techniques will be incorporated into the program. Participants will also have the option to join a weekly group telehealth call via Skype for Business. The main researcher, a physiotherapist specialized in PA counselling in mental health, will lead the discussion and provide further education on the same weekly topic as the Facebook group for approximately 20-30 min. To encourage participation, there will be two telehealth group calls per week and participants can join either. Participants will be able to join in on the discussion, share their experiences, and ask questions. Participants allocated to the control group will be assigned to a waiting list and enter the Facebook Group after the last follow-up assessment. The control group will receive the same content but there will be no telehealth discussion calls.

Table 1. Content of the on-line intervention. Week Content

1. Welcome and introductions.
2. Goal setting and self-monitoring.
3. Sedentary behaviour and recommendation
4. Physical and mental health benefits of PA.
5. Barriers and motivations.
6. Mental contrasting.
7. Support
8. Aerobic exercise.
9. Resistance exercise.
10. Review program / congratulations.

Data analysis:

Statistical analyses will be run using IBM SPSS statistics version 27. Data will be tested for normality with the Shapiro-Wilks test. Differences in baseline characteristics between the two groups will be analysed by means of independent-samples t-tests or Mann Whitney U tests when appropriate for continuous variables, and Chi-square test for categorical variables. Pre-specified intention-to-treat analysis will consider participants randomly assigned to each group for inclusion in the analysis, using the base-line characteristics of non-completers to compare with participants who complete all follow-up assessments. Multivariate analysis of variance will be used to explore between-group differences (standard mean difference and 95% confidence intervals) immediately post-intervention and at 3-month follow-up for all outcome measures. Cohen's d will be used as an estimate of the effect size. Mediation analysis will be carried out in 3 steps. First, effects of the intervention on autonomous motivation and perceived social support (potential mediators) will be tested by regressing both variables into the treatment condition. Second, associations between changes in potential mediators and changes in PA levels and mental health outcomes will be assessed by regressing PA levels and mental health outcomes into treatment condition and potential mediators. Third, indirect effect will be estimated and tested for statistical significance by means of the Sobel test.

Qualitative analysis will be based on an Interpretative Phenomenological Approach. QRS Internationals' NVivo 12 software will be used to store and code the inductive qualitative data gathered from the focus groups. Interviews will be recorded and transcribed verbatim, and sent back to the participant to check veracity. In order to identify, analyse, and report patterns within data, thematic analysis will be used. The steps for thematic analysis are: 1) familiarisation with data, 2) generation of initial codes, 3) searching for themes, 4) reviewing the themes, 5) defining and naming the themes, and 6) producing the report. Trustworthiness will be ensured by team meetings to discuss the data. A research assistant will take the role of observer in the focus-groups and assist the main researcher with data collection and non-verbal observations.

Compliance and acceptability:

Will be defined by usage of the Facebook group (manual calculation of the sum of posts, likes and comments), and participant retention (completion of questionnaires and retention in programme). Acceptability will be assessed immediately post-intervention using the 14-item feasibility and acceptability questionnaire that has been used previously to measure participant responses to a private Facebook group.

Ethical considerations:

All participants will receive information concerning the purpose of the study, being properly stated in a consent form in Dutch. The protocol, patient data management plan, and consent form will be sent to the local KU Leuven Ethical Committee, and registered at clinical trial center (CTC) UZ Leuven prior to the start of the trial. To avoid potential loss of confidentiality, data collected will be anonymized and de-identified immediately after its collection. For qualitative focus groups, participants' names will be coded in a password-secured file by the main researcher. Participation in all studies is voluntary and participants will be able to withdraw at any time without any consequence or prejudice. Participation in the intervention study will not be reimbursed since monetary profit is a form of external motivation which might affect the outcomes of the intervention. Flyers showcasing the obtained results will be sent to the involved associations for their dissemination.

Participation in these studies has little to no associated risks. Participants that are confronted with strong emotions when filling in the surveys will be directed to local psychological services. There will be no direct human contact, implying no COVID-19 infection risk. All data collection will be carried out on-line, and post PA recommendations will be adapted to current local restrictions and recommendations (consulted in https://www.info-coronavirus.be/en/faq/).

Facebook group will be private and hidden for anyone not involved in the intervention. Participants will be encouraged to make anonymous posts when discussing sensible topics in the Facebook group. Anonymous posts are seen by every member of the group but only the group administrator will know the identity of the person posting it. Additionally, participants will have to sign a confidentiality clause in order to enter the group. During telehealth calls and focus groups, only the first name of the participants will be used.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Physically inactive (less than 150 minutes of moderate to vigorous physical activity per week)
* Active as a firefighter
* At least mild symptoms of depression, anxiety or stress according to the DASS-21

Exclusion Criteria:

* Acute suicide ideation
* Unfit to engage in physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-11 (Estimated); Primary Completion 2022-08-23 (Estimated); Study Completion 2022-08-23 (Estimated)

PRIMARY OUTCOMES:
Simple Physical Activity Questionnaire. Changes in Physical Activity levels | Baseline, immediately after intervention, at 3 months follow-up
  5-item clinical tool to assess physical activity levels among populations at high risk for physical inactivity.
PTSD checklist for the DSM-5. Changes in PTSD symptoms. | Baseline, immediately after intervention, at 3 months follow-up
  A self-report assessment tool that measures symptoms of post-traumatic stress according to the DSM-5 during the past month with the aim of monitoring symptom change, screening individuals for PTSD, or making a provisional PTSD diagnosis. Higher scores imply more severity, ranging from 0 to 80.

SECONDARY OUTCOMES:
Behavioural Regulation for Exercise, Third Edition. Changes in quality of motivation | Baseline, immediately after intervention, at 3 months follow-up
  Evaluates different aspects of motivation towards exercise which includes the items for integrated regulation.
Alcohol Use Disorders Identification Test. Changes in Alcohol use. | Baseline, immediately after intervention, at 3 months follow-up
  The AUDIT is an assessment tool developed by the World Health Organisation (WHO) and used for evaluating risky alcohol consumption patterns.
Social Support for Exercise Behaviours Scale. Changes in Social Support. | Baseline, immediately after intervention, at 3 months follow-up
  a self-report scale designed to assess social support for exercise across 3 domains, namely Family support: participation and involvement; Family support: rewards and punishments; and Friends support: exercising together. Higher scores mean higher social support,
Pittsburgh Sleep Quality Index. Changes in Sleep Quality. | Baseline, immediately after intervention, at 3 months follow-up
  The PSQI is a self-report assessment tool that measures sleep quality during the previous month.
The Depression and Anxiety Stress Scale - 21. Changes in symptoms of depression, anxiety, and stress. | Baseline, immediately after intervention, at 3 months follow-up
  The DASS-21 is a self-report assessment tool that measures symptoms of depression, anxiety, and stress over the past week. Scores range from 0 to 63, with higher scores meaning more severe symptoms.
WHO-5 Well-being - index. Changes in quality of life | Baseline, immediately after intervention, at 3 months follow-up
  a self-report assessment tool that measures general well-being over the past 2 weeks. It contains 5 questions rated on a 6-point Likert scale ranging from 0 (at no time) to 5 (all of the time), with higher scores indicating better well-being.
Global Psychotrauma Screen. Changes in trauma symptoms. | Baseline, immediately after intervention, at 3 months follow-up
  The GPS is an assessment tool designed for screening for a range of trauma-related psychological problems, as well as for risk of protective factors. It consists of 22 yes / no questions.

CONTACTS AND LOCATIONS:
Overall Officials: Davy Vancampfort, dr, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aertgeerts B, Buntinx F, Ansoms S, Fevery J. Questionnaires are better than laboratory tests to screen for current alcohol abuse or dependence in a male inpatient population. Acta Clin Belg. 2002 Sep-Oct;57(5):241-9. doi: 10.1179/acb.2002.048. PMID 12534130
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA: Author.
- [Background] Anderson ES, Wojcik JR, Winett RA, Williams DM. Social-cognitive determinants of physical activity: the influence of social support, self-efficacy, outcome expectations, and self-regulation among participants in a church-based health promotion study. Health Psychol. 2006 Jul;25(4):510-20. doi: 10.1037/0278-6133.25.4.510. PMID 16846326
- [Background] Ashdown-Franks G, Sabiston CM, Stubbs B. The evidence for physical activity in the management of major mental illnesses: a concise overview to inform busy clinicians' practice and guide policy. Curr Opin Psychiatry. 2019 Sep;32(5):375-380. doi: 10.1097/YCO.0000000000000526. PMID 31145143
- [Background] Ashdown-Franks G, Firth J, Carney R, Carvalho AF, Hallgren M, Koyanagi A, Rosenbaum S, Schuch FB, Smith L, Solmi M, Vancampfort D, Stubbs B. Exercise as Medicine for Mental and Substance Use Disorders: A Meta-review of the Benefits for Neuropsychiatric and Cognitive Outcomes. Sports Med. 2020 Jan;50(1):151-170. doi: 10.1007/s40279-019-01187-6. PMID 31541410
- [Background] Babor, T. F., Higgins-Biddle, J. C., Saunders, J. B., & Monteiro, M. G. (2001). The alcohol use disorders identification test.
- [Background] Berger W, Coutinho ES, Figueira I, Marques-Portella C, Luz MP, Neylan TC, Marmar CR, Mendlowicz MV. Rescuers at risk: a systematic review and meta-regression analysis of the worldwide current prevalence and correlates of PTSD in rescue workers. Soc Psychiatry Psychiatr Epidemiol. 2012 Jun;47(6):1001-11. doi: 10.1007/s00127-011-0408-2. Epub 2011 Jun 18. PMID 21681455
- [Background] Bisson JI, Berliner L, Cloitre M, Forbes D, Jensen TK, Lewis C, Monson CM, Olff M, Pilling S, Riggs DS, Roberts NP, Shapiro F. The International Society for Traumatic Stress Studies New Guidelines for the Prevention and Treatment of Posttraumatic Stress Disorder: Methodology and Development Process. J Trauma Stress. 2019 Aug;32(4):475-483. doi: 10.1002/jts.22421. Epub 2019 Jul 8. PMID 31283056
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative research in psychology, 3(2), 77-101.
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cid L, Monteiro D, Teixeira D, Teques P, Alves S, Moutao J, Silva M, Palmeira A. The Behavioral Regulation in Exercise Questionnaire (BREQ-3) Portuguese-Version: Evidence of Reliability, Validity and Invariance Across Gender. Front Psychol. 2018 Oct 11;9:1940. doi: 10.3389/fpsyg.2018.01940. eCollection 2018. PMID 30364299
- [Background] Hall KS, Hoerster KD, Yancy WS Jr. Post-traumatic stress disorder, physical activity, and eating behaviors. Epidemiol Rev. 2015;37:103-15. doi: 10.1093/epirev/mxu011. Epub 2015 Jan 16. PMID 25595169
- [Background] Ehring T, Zetsche U, Weidacker K, Wahl K, Schonfeld S, Ehlers A. The Perseverative Thinking Questionnaire (PTQ): validation of a content-independent measure of repetitive negative thinking. J Behav Ther Exp Psychiatry. 2011 Jun;42(2):225-32. doi: 10.1016/j.jbtep.2010.12.003. Epub 2010 Dec 21. PMID 21315886
- [Background] Jones S, Agud K, McSweeney J. Barriers and Facilitators to Seeking Mental Health Care Among First Responders: "Removing the Darkness". J Am Psychiatr Nurses Assoc. 2020 Jan/Feb;26(1):43-54. doi: 10.1177/1078390319871997. Epub 2019 Sep 11. PMID 31509058
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Firth J, Solmi M, Wootton RE, Vancampfort D, Schuch FB, Hoare E, Gilbody S, Torous J, Teasdale SB, Jackson SE, Smith L, Eaton M, Jacka FN, Veronese N, Marx W, Ashdown-Franks G, Siskind D, Sarris J, Rosenbaum S, Carvalho AF, Stubbs B. A meta-review of "lifestyle psychiatry": the role of exercise, smoking, diet and sleep in the prevention and treatment of mental disorders. World Psychiatry. 2020 Oct;19(3):360-380. doi: 10.1002/wps.20773. PMID 32931092
- [Background] Firth J, Ward PB, Stubbs B. Editorial: Lifestyle Psychiatry. Front Psychiatry. 2019 Aug 26;10:597. doi: 10.3389/fpsyt.2019.00597. eCollection 2019. No abstract available. PMID 31507466
- [Background] Gomez, F. (2016). A guide to the depression, anxiety and stress scale (DASS 21). Central and Eastern Sydney primary health networks.
- [Background] Gonzalez-Cutre D, Sicilia A, Fernandez A. [Toward a deeper understanding of motivation towards exercise: measurement of integrated regulation in the Spanish context]. Psicothema. 2010 Nov;22(4):841-7. Spanish. PMID 21044522
- [Background] Greenwood JL, Joy EA, Stanford JB. The Physical Activity Vital Sign: a primary care tool to guide counseling for obesity. J Phys Act Health. 2010 Sep;7(5):571-6. doi: 10.1123/jpah.7.5.571. PMID 20864751
- [Background] Hagger MS, Hardcastle SJ, Chater A, Mallett C, Pal S, Chatzisarantis NL. Autonomous and controlled motivational regulations for multiple health-related behaviors: between- and within-participants analyses. Health Psychol Behav Med. 2014 Jan 1;2(1):565-601. doi: 10.1080/21642850.2014.912945. Epub 2014 Apr 30. PMID 25750803
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Hinz A, Glaesmer H, Brahler E, Loffler M, Engel C, Enzenbach C, Hegerl U, Sander C. Sleep quality in the general population: psychometric properties of the Pittsburgh Sleep Quality Index, derived from a German community sample of 9284 people. Sleep Med. 2017 Feb;30:57-63. doi: 10.1016/j.sleep.2016.03.008. Epub 2016 May 4. PMID 28215264
- [Background] Kaniasty, K. (2012). Predicting social psychological well-being following trauma: The role of postdisaster social support. Psychological Trauma: Theory, Research, Practice, and Policy, 4(1), 22. 19
- [Background] Kelley GA, Kelley KS. Exercise and sleep: a systematic review of previous meta-analyses. J Evid Based Med. 2017 Feb;10(1):26-36. doi: 10.1111/jebm.12236. PMID 28276627
- [Background] Kroll T, Morris J. Challenges and opportunities in using mixed method designs in rehabilitation research. Arch Phys Med Rehabil. 2009 Nov;90(11 Suppl):S11-6. doi: 10.1016/j.apmr.2009.04.023. PMID 19892069
- [Background] Kim JE, Dager SR, Jeong HS, Ma J, Park S, Kim J, Choi Y, Lee SL, Kang I, Ha E, Cho HB, Lee S, Kim EJ, Yoon S, Lyoo IK. Firefighters, posttraumatic stress disorder, and barriers to treatment: Results from a nationwide total population survey. PLoS One. 2018 Jan 5;13(1):e0190630. doi: 10.1371/journal.pone.0190630. eCollection 2018. PMID 29304155
- [Background] Lara-Cabrera ML, Mundal IP, De Las Cuevas C. Patient-reported well-being: psychometric properties of the world health organization well-being index in specialised community mental health settings. Psychiatry Res. 2020 Sep;291:113268. doi: 10.1016/j.psychres.2020.113268. Epub 2020 Jun 30. PMID 32629296
- [Background] Lardier DT, Coakley KE, Holladay KR, Amorim FT, Zuhl MN. Exercise as a Useful Intervention to Reduce Alcohol Consumption and Improve Physical Fitness in Individuals With Alcohol Use Disorder: A Systematic Review and Meta-Analysis. Front Psychol. 2021 Jul 7;12:675285. doi: 10.3389/fpsyg.2021.675285. eCollection 2021. PMID 34305729
- [Background] Long, N., Readdy, T., & Raabe, J. (2014). What motivates firefighters to exercise? A mixed-methods investigation of self-determination theory constructs and exercise behavior. Sport, Exercise, and Performance Psychology, 3(3), 203.
- [Background] Markland, D., & Tobin, V. (2004). A modification to the behavioural regulation in exercise questionnaire to include an assessment of amotivation. Journal of Sport and Exercise Psychology, 26(2), 191-196.
- [Background] Martin ZT, Schlaff RA, Hemenway JK, Coulter JR, Knous JL, Lowry JE, Ode JJ. Cardiovascular Disease Risk Factors and Physical Fitness in Volunteer Firefighters. Int J Exerc Sci. 2019 May 1;12(2):764-776. doi: 10.70252/MGCY6653. eCollection 2019. PMID 31156744
- [Background] McKeon G, Steel Z, Wells R, Newby JM, Hadzi-Pavlovic D, Vancampfort D, Rosenbaum S. Mental health informed physical activity for first responders and their support partner: a protocol for a stepped-wedge evaluation of an online, codesigned intervention. BMJ Open. 2019 Sep 11;9(9):e030668. doi: 10.1136/bmjopen-2019-030668. PMID 31511290
- [Background] McKeon, G., Wells, R., Steel, Z., Moseley, V., & Rosenbaum, S. (2020). Self-Reported Physical and Mental Health of Informal Caregivers of Emergency Service Workers. Journal of Loss and Trauma, 1-12.
- [Background] McKim, C. A. (2017). The value of mixed methods research: A mixed methods study. Journal of Mixed Methods Research, 11(2), 202-222.
- [Background] Moran, J., Kelly, G., Haberlin, C., Mockler, D., & Broderick, J. (2018). The use of eHealth to promote physical activity in people with mental health conditions: a systematic review. HRB Open Research, 1, 5.
- [Background] Naslund JA, Aschbrenner KA, Marsch LA, McHugo GJ, Bartels SJ. Facebook for Supporting a Lifestyle Intervention for People with Major Depressive Disorder, Bipolar Disorder, and Schizophrenia: an Exploratory Study. Psychiatr Q. 2018 Mar;89(1):81-94. doi: 10.1007/s11126-017-9512-0. PMID 28470468
- [Background] Palinkas LA, Horwitz SM, Chamberlain P, Hurlburt MS, Landsverk J. Mixed-methods designs in mental health services research: a review. Psychiatr Serv. 2011 Mar;62(3):255-63. doi: 10.1176/ps.62.3.pss6203_0255. PMID 21363896
- [Background] Rauscher L, Greenfield BH. Advancements in contemporary physical therapy research: use of mixed methods designs. Phys Ther. 2009 Jan;89(1):91-100. doi: 10.2522/ptj.20070236. Epub 2008 Nov 13. PMID 19008328
- [Background] Rhodes RE, Pfaeffli LA. Mediators of physical activity behaviour change among adult non-clinical populations: a review update. Int J Behav Nutr Phys Act. 2010 May 11;7:37. doi: 10.1186/1479-5868-7-37. PMID 20459781
- [Background] Rosenbaum S, Morell R, Abdel-Baki A, Ahmadpanah M, Anilkumar TV, Baie L, Bauman A, Bender S, Boyan Han J, Brand S, Bratland-Sanda S, Bueno-Antequera J, Camaz Deslandes A, Carneiro L, Carraro A, Castaneda CP, Castro Monteiro F, Chapman J, Chau JY, Chen LJ, Chvatalova B, Chwastiak L, Corretti G, Dillon M, Douglas C, Egger ST, Gaughran F, Gerber M, Gobbi E, Gould K, Hatzinger M, Holsboer-Trachsler E, Hoodbhoy Z, Imboden C, Indu PS, Iqbal R, Jesus-Moraleida FR, Kondo S, Ku PW, Lederman O, Lee EHM, Malchow B, Matthews E, Mazur P, Meneghelli A, Mian A, Morseth B, Munguia-Izquierdo D, Nyboe L, O'Donoghue B, Perram A, Richards J, Romain AJ, Romaniuk M, Sadeghi Bahmani D, Sarno M, Schuch F, Schweinfurth N, Stubbs B, Uwakwe R, Van Damme T, Van Der Stouwe E, Vancampfort D, Vetter S, Waterreus A, Ward PB. Assessing physical activity in people with mental illness: 23-country reliability and validity of the simple physical activity questionnaire (SIMPAQ). BMC Psychiatry. 2020 Mar 6;20(1):108. doi: 10.1186/s12888-020-2473-0. PMID 32143714
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Schuch FB, Vancampfort D, Richards J, Rosenbaum S, Ward PB, Stubbs B. Exercise as a treatment for depression: A meta-analysis adjusting for publication bias. J Psychiatr Res. 2016 Jun;77:42-51. doi: 10.1016/j.jpsychires.2016.02.023. Epub 2016 Mar 4. PMID 26978184
- [Background] Schnyder U, Schafer I, Aakvaag HF, Ajdukovic D, Bakker A, Bisson JI, Brewer D, Cloitre M, Dyb GA, Frewen P, Lanza J, Le Brocque R, Lueger-Schuster B, Mwiti GK, Oe M, Rosner R, Schellong J, Shigemura J, Wu K, Olff M. The global collaboration on traumatic stress. Eur J Psychotraumatol. 2017 Nov 30;8(sup7):1403257. doi: 10.1080/20008198.2017.1403257. eCollection 2017. PMID 29435201
- [Background] Schuch FB, Stubbs B. The Role of Exercise in Preventing and Treating Depression. Curr Sports Med Rep. 2019 Aug;18(8):299-304. doi: 10.1249/JSR.0000000000000620. PMID 31389872
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. Trials. 2010 Mar 24;11:32. doi: 10.1186/1745-6215-11-32. PMID 20334632
- [Background] Stubbs B, Vancampfort D, Rosenbaum S, Firth J, Cosco T, Veronese N, Salum GA, Schuch FB. An examination of the anxiolytic effects of exercise for people with anxiety and stress-related disorders: A meta-analysis. Psychiatry Res. 2017 Mar;249:102-108. doi: 10.1016/j.psychres.2016.12.020. Epub 2017 Jan 6. PMID 28088704
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Tremblay MS, Aubert S, Barnes JD, Saunders TJ, Carson V, Latimer-Cheung AE, Chastin SFM, Altenburg TM, Chinapaw MJM; SBRN Terminology Consensus Project Participants. Sedentary Behavior Research Network (SBRN) - Terminology Consensus Project process and outcome. Int J Behav Nutr Phys Act. 2017 Jun 10;14(1):75. doi: 10.1186/s12966-017-0525-8. PMID 28599680
- [Background] Tuohy D, Cooney A, Dowling M, Murphy K, Sixsmith J. An overview of interpretive phenomenology as a research methodology. Nurse Res. 2013 Jul;20(6):17-20. doi: 10.7748/nr2013.07.20.6.17.e315. PMID 23909107
- [Background] Wilson, P. M., Rodgers, W. M., Loitz, C. C., & Scime, G. (2006). "It's Who I Am… Really! 'The importance of integrated regulation in exercise contexts 1. Journal of Applied Biobehavioral Research, 11(2), 79-104.
- [Background] Wortmann JH, Jordan AH, Weathers FW, Resick PA, Dondanville KA, Hall-Clark B, Foa EB, Young-McCaughan S, Yarvis JS, Hembree EA, Mintz J, Peterson AL, Litz BT. Psychometric analysis of the PTSD Checklist-5 (PCL-5) among treatment-seeking military service members. Psychol Assess. 2016 Nov;28(11):1392-1403. doi: 10.1037/pas0000260. Epub 2016 Jan 11. PMID 26751087
- [Background] Vancampfort D, Sanchez CPR, Hallgren M, Schuch F, Firth J, Rosenbaum S, Van Damme T, Stubbs B. Dropout from exercise randomized controlled trials among people with anxiety and stress-related disorders: A meta-analysis and meta-regression. J Affect Disord. 2021 Mar 1;282:996-1004. doi: 10.1016/j.jad.2021.01.003. Epub 2021 Jan 6. PMID 33601745
- [Background] Zegel M, Lebeaut A, Healy N, Tran JK, Vujanovic AA. Mental Health Correlates of Probable Posttraumatic Stress Disorder, Probable Alcohol Use Disorder, and Their Co-Occurrence among Firefighters. Behav Modif. 2022 Mar;46(2):395-421. doi: 10.1177/01454455211033517. Epub 2021 Jul 29. PMID 34323099
- [Background] Ramos-Sanchez CP, Schuch FB, Seedat S, Louw QA, Stubbs B, Rosenbaum S, Firth J, van Winkel R, Vancampfort D. The anxiolytic effects of exercise for people with anxiety and related disorders: An update of the available meta-analytic evidence. Psychiatry Res. 2021 Aug;302:114046. doi: 10.1016/j.psychres.2021.114046. Epub 2021 Jun 11. PMID 34126464
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232